CLINICAL TRIAL: NCT02258503
Title: Impact of the Use of the Scale ALGOPLUS® on the Prescriptions of Analgesics in Emergency Department on Patients of 75 Years Old or More
Acronym: DOLEVA75
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0211
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: Numerical scale; Pain in elderly patients admitted in emergency department
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- numerical scale: Evaluation of the pain of elderly patient admitted in the emergency department by numerical scale and then taken care according to the usual practice of the emergency department.
  Interventions: Other: pain in elderly patients
- algoplus scale: Evaluation of the pain of elderly patient admitted in the emergency department by numerical scale and by Algoplus® scale then taken care according to the usual practice of the emergency department.
  Interventions: Other: pain in elderly patients

INTERVENTIONS:
Other: pain in elderly patients

SUMMARY:
The pain of the elderly is even often unrecognized or trivialized and ignored in spite of its big frequency: the chronic pain affects 50 % of the elderly living at home, 49 to 83 % of those living in institution and 80 % of this population at the end of life.

So in the elderly, the noxious character of the pain is more pregnant than at the young adult. The echo on the acts of the everyday life is fast, the activities decrease, coming to deteriorate the isolation and the dependence: the echo on the psychic state is frequent and the pain is a part of the cause of a confusional state. Finally, the presence of a pain distorts considerably the quality of life and can modify the state general as the desire of life.

The evaluation of the pain appeals to the same strategy as to the younger subject but with some specificities, related more to the pathologies associated with the ageing than with the real age. For that purpose, the investigators have first of all scale of self-assessment as the numerical scale which is adapted to estimate the acute and chronic pains but this scale presents a bias because, certain patients do not express spontaneously their pain and this one must be attentively looked for in case of modification of behavior.

So scales of hetero-evaluation were elaborated to solve the difficulties of detection and to care the pain of the elderly. One of these is the scale Algoplus® (5 items which allow within one minute a good quality evaluation whatever is the place of care) whose objective is the observation of the behavioral changes caused by the acute pain in elderly having communication disorders.

Due to the demographic evolution, emergency departments are more and more frequently a place of consultation of the elderly. Indeed, the elderly represent approximately 10 to 20 % of all the passages in emergency department and 50 % of the patients hospitalized during the passage in the reception of Emergency department are elderly. Elderly care is difficult for a certain number of reasons (vulnerability, accumulation of pathologies and treatments). So, in this context, the evaluation of the presence of pain and its care are difficult in particular at the elderly with communication disorders.

In a preliminary study in the emergency department of the Hospital of Clermont-Ferrand, on 700 patients of more than 75 years old admitted in April 2012, 32 % had a prescription of analgesic while 13 % only had a real quotation of the pain.

The aim of the investigators study is to analyze if the systematic introduction of the scale Algoplus® in the evaluation of elderly during its entrance to emergency department could modify the prescription of analgesic.

DETAILED DESCRIPTION:
First period of the study :

Evaluation of the pain of elderly patient admitted in the emergency department by numerical scale and then taken care according to the usual practice of the emergency department.

A Clinical Research Associate will collect the quotation of pain by numerical scale and the analgesics treatments prescribed and their posology and route of administration.

This data collection must be realized for 100 elderly patients of 75 or more years old admitted the Emergency department during one month.

Training period :

Training of the emergency physicians in the use of the Algoplus® scale.

Second period of the study :

Evaluation of the pain of elderly patient admitted in the emergency department by numerical scale and by Algoplus® scale then taken care according to the usual practice of the emergency department.

A Clinical Research Associate will collect the quotation of pain by numerical scale and by Algoplus® scale and the analgesics treatments prescribed and their posology and route of administration.

This data collection must be realized for 100 elderly patients of 75 or more years old admitted the Emergency department during one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in emergency department for any pathologies,
* Patients of 75 or more years old

Exclusion Criteria:

* Patients of less than 75 years.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Collection of the rate of prescription of analgesic treatments | at day 1

SECONDARY OUTCOMES:
Collection of the score of quotation of pain by numerical scale (score from 0 to 10) | at day 1
Collection of prescription of analgesic | at day 1
Collection of the prescription of analgesic by class according to the scale of the WHO | at day 1
Collection of the score of the scale Algoplus® | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France